CLINICAL TRIAL: NCT07093307
Title: Using a Docudrama Intervention to Increase Repeat Donation Among First-time Blood Donors in Ghana: a Pilot Cluster Randomized, Pragmatic Type 1 Effectiveness- Implementation Hybrid Trial
Brief Title: Docudrama for Blood Donation in Ghana (DDID)
Acronym: DDID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Syracuse University (Other); National Blood Service Ghana (Other); University of Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B11; 4UH3HL151599-03 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Blood Donation
Keywords: Docudrama

STUDY DESIGN:
Intervention Model Description: Cluster randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docudrama (Experimental)
  Interventions: Behavioral: Docudrama
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Docudrama — Participants at docudrama sites will watch a 30-minute docudrama (two episodes of 15 minutes each) immediately after blood donation while waiting to recover and to be refreshed.
  Arms: Docudrama
Behavioral: Control — Participants randomized at control sites will receive the standard NBSG communications for blood donors: 1) a "thank you" phone call and 2) and a reminder phone call two-weeks prior to when they are due for their next blood donation.
  Arms: Control

SUMMARY:
A cluster pilot RCT to evaluate the effectiveness of the docudrama compared to a control group (usual engagement with blood services) on repeat blood donation attempts among first-time blood donors. Secondary outcomes will be blood donor retention, attitudes, subjective norms, perceived behavioral control and intention as potential mediators of blood donation behavior among first-time blood donors. The cluster pilot RCT will have two arms: 1) docudrama and 2) control. Randomization will stratify by the type of site: mobile versus fixed. Each participant in the docudrama arm will receive the intervention one time immediately after blood donation. Participants in both the docudrama arm and control arm will receive standard blood donor communications and will be followed for six months. Actualized blood donation is possible every four months using NBSG guidelines; however, blood donation sessions may not occur at the blood donation sites until six months. Return blood donation attempts will be evaluated using the Southern Zonal Blood Center (SZBC) records (primary outcome) and participant self-report (secondary outcome) at six months. Secondary measures will be evaluated at baseline and six months from enrollment. The duration of the study will be 11 months, allowing for five months to achieve enrollment goals and six months of follow-up for the last individual enrolled.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years-old
* First-time whole blood donor with the SZBC of the NBSG
* Eligible to donate again at the time of eligibility confirmation
* Consent to participate
* Has a valid contact phone number or access to a valid contact phone number
* Understands one of English, Twi, or Ga
* Be willing to watch a docudrama on blood donation

Exclusion Criteria:

* History of more than one lifetime whole blood donation (with any blood center)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a verified repeat blood donation attempt | Within 6 months after randomization
  Self-report of a blood donation attempt at the 6 month follow-up phone call using a questionnaire that is administered by study research staff over the phone. Self-reported attempts are then verified using the National Blood Services Ghana (NBSG) national blood donation database.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Zonal Blood Centre, National Blood Service Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided